CLINICAL TRIAL: NCT01124643
Title: An Open-label Extension of Study TKT028 Evaluating Safety and Clinical Outcomes of Replagal® Enzyme Replacement Therapy Administered to Adult Patients With Fabry Disease
Brief Title: Extension Study of TKT028 Evaluating Safety and Clinical Outcomes of Replagal® in Adult Patients With Fabry Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGT-REP-060; 2009-015985-75 (EudraCT Number)
Record Dates: First submitted 2010-04-23; First posted 2010-05-17 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Fabry Disease
Keywords: Agalsidase alfa; Alpha-Galactosidase; Replagal; Enzyme Replacement Therapy
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase alfa; alpha-Galactosidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Replagal 0.2 mg/kg EOW (Experimental): Intravenous, 0.2mg/kg EOW
  Interventions: Biological: Replagal

INTERVENTIONS:
Biological: Replagal — 0.2 mg/kg administered intravenously [IV] every other week
  Other Names: algalsidase alfa; alpha-Galactosidase; DRX005B

SUMMARY:
This study will evaluate safety and clinical outcomes of treatment with Replagal in adult participants with Fabry disease who have completed Study TKT028 (NCT00864851).

DETAILED DESCRIPTION:
HGT-REP-060 was designed to provide participants who participated in TKT028 an additional 52 weeks of treatment with Replagal at the standard dose of 0.2 milligram per kilogram (mg/kg) every other week (EOW) to assess the effect of continued Replagal therapy on long-term safety and clinical outcomes for this participant population.

ELIGIBILITY:
Inclusion Criteria:

* Complete all study requirements and assessments for Study TKT028 less than 30 days (+/- 7 days) prior to the first dose in this extension protocol
* Voluntarily signed an Institutional Review Board/Independent Ethics Committee- approved informed consent form after all relevant aspects of the study have been explained and discussed.
* Has received and tolerated at least 80% of the total planned Replagal infusions in Study TKT028
* Female participants of child-bearing potential must agree to use a medically acceptable method of contraception at all times during the study and must have a negative pregnancy test at the time of study entry and as required throughout participation in study

Exclusion Criteria:

* Has received treatment with any investigational drug (other than Replagal) or device within 30 days prior to study entry.
* Is unable to comply with the protocol, (eg, is unable to return for safety evaluations, or is otherwise unlikely to complete the study), as determined by the Investigator
* Has a positive test for hepatitis B surface antigen (HBsAg), hepatitis C(HCV) antibody, or human immunodeficiency virus (HIV) antibody
* Is pregnant or lactating
* Is morbidly obese, defined as body mass index (BMI) >39 kg/m2
* Has any safety or medical issues, as assessed by the Investigator, that contraindicate participation in the study (eg, has experienced an adverse reaction to treatment with Replagal or has a known hypersensitivity to any of the components of Replagal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-04-13 (Actual); Primary Completion 2013-07-08 (Actual); Study Completion 2013-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- United States (2):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - O&O Alpan LLC, Fairfax, Virginia
- The Royal Melbourne Hospital, Parkville, Australia
- 1st School of Medicine Charles University, Prague, Czechia
- Turku University Central Hospital, Turku, Finland
- Poland (2):
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Instytut Kardiologii, I Klinika Choroby Wiencowej, Warsaw
- General Hospital Slovenj Gradec, Slovenj Gradec, Slovenia
- Salford Royal NHS Foundation Trust, Salford, England, United Kingdom

REFERENCES:
- [Result] Golan L, Goker-Alpan O, Holida M, Kantola I, Klopotowski M, Kuusisto J, Linhart A, Musial J, Nicholls K, Gonzalez-Rodriguez D, Sharma R, Vujkovac B, Chang P, Wijatyk A. Evaluation of the efficacy and safety of three dosing regimens of agalsidase alfa enzyme replacement therapy in adults with Fabry disease. Drug Des Devel Ther. 2015 Jul 8;9:3435-44. doi: 10.2147/DDDT.S80928. eCollection 2015. PMID 26185417

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening details: Thirty-five of the 40 subjects who completed the parent study (Study TKT028 [NCT00864851]) were enrolled in this extension study.
Groups:
- Replagal® (0.2 mg/kg): Replagal 0.2 milligram per kilogram (mg/kg) intravenously (IV), every other week (EOW).
Period: Overall Study
Arm/Group | Replagal® (0.2 mg/kg)
Started | 35
Completed | 34
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Replagal® (0.2 mg/kg): Replagal 0.2 mg/kg IV, EOW
Arm/Group | Replagal® (0.2 mg/kg)
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.3 (9.86)
Age, Customized [Count of Participants; unit: Participants] — Age at time of consent
  Participants
    >=65 years | 3
    Between 18 and 65 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 19
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRALIA | 2
  CZECH REPUBLIC | 5
  FINLAND | 5
  POLAND | 13
  SLOVENIA | 4
  UNITED KINGDOM | 3
  UNITED STATES | 3
Left Ventricular Mass Indexed to Height (LVMI) [Mean (Standard Deviation); unit: gram per meter to the power 2.7(g/m^2.7)] — Number of participants analyzed for this baseline characteristic was 33
  gram per meter to the power 2.7(g/m^2.7) | 81.18 (32.13)
Maximal Oxygen Consumption (VO2max) [Mean (Standard Deviation); unit: milliliter/minute/kilogram (mL/min/kg)] — Number of participants analyzed for this baseline characteristic was 32
  milliliter/minute/kilogram (mL/min/kg) | 20.2 (6.73)
Distance Walked in 6-Minute Walk Test (6MWT) [Mean (Standard Deviation); unit: meters] — Number of participants analyzed for this baseline characteristic was 34
  meters | 515.5 (144.13)
Minnesota Living with Heart Failure Questionnaire (MLHF-Q) Summary Score [Mean (Standard Deviation); unit: units on a scale] — The MLHF-Q contains 21 questions with answers ranging from 0 (no) to 5 (very much). The final score ( 0 to 105) is the sum of the points for the 21 questions. A higher score indicates a worse quality of life.
  units on a scale | 26.5 (26.95)
New York Heart Association (NYHA) Functional Class [Count of Participants; unit: Participants] — Class I = No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea Class II = Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea Class III = Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea Class IV = Unable to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. If any physical activity is undertaken, discomfort is increased
  Participants
    Class I (Very Mild) | 21
    Class II (Mild) | 13
    Class III (Moderate) | 1
    Class IV (Severe) | 0
Plasma Gb3 (globotriaosylceramide) [Mean (Standard Deviation); unit: nanomoles per milliliter (nmol/mL)] | 4.35 (2.51)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: (mL/min/1.73m^2)] | 77.60 (26.12)
Albumin-to-Creatinine (A/Cr) Ratio [Mean (Standard Deviation); unit: Ratio] — Number of participants analyzed for this baseline characteristic was 33
  Ratio | 284.1 (712.90)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Left Ventricular Mass Indexed to Height (LVMI)
Time Frame: Baseline to 12 months
Population: The Intent-to-Treat (ITT) participant population in this study was defined as all participants who provided informed consent and received study drug. Participants who did not have left ventricular hypertrophy were not included in this analysis.
Measure: Mean (Standard Deviation); unit: g/m^2.7
Arm/Group | Replagal® (0.2 mg/kg)
Number analyzed (Participants) | 32
g/m^2.7 | -0.75 (13.46)

2. Secondary Outcome: Change From Baseline in Maximal Oxygen Consumption (VO2max) at Peak Exercise
Time Frame: Baseline to 12 months
Population: ITT population. Test was not done or test was not valid for all participants.
Measure: Mean (Standard Deviation); unit: (mL/min/kg)
Arm/Group | Replagal® (0.2 mg/kg)
Number analyzed (Participants) | 28
(mL/min/kg) | -0.7 (3.11)

3. Secondary Outcome: Change From Baseline in Distance Walked in 6- Minute Walk Test (6MWT)
Time Frame: Baseline to 12 months
Population: ITT population. Test was not done or test was not valid for all participants.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Replagal® (0.2 mg/kg)
Number analyzed (Participants) | 32
meters | -11.2 (83.99)

4. Secondary Outcome: Change From Baseline in the Minnesota Living With Heart Failure Questionnaire (MLHF- Q)
Description: The MLHF-Q contains 21 questions with answers ranging from 0 (no) to 5 (very much). The final score ( 0 to 105) is the sum of the points for the 21 questions. A higher score indicates a worse quality of life.
Time Frame: Baseline to 12 months
Population: ITT population. Number of participants analyzed signifies participants evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Replagal® (0.2 mg/kg)
Number analyzed (Participants) | 34
units on a scale | 6.0 (19.31)

5. Secondary Outcome: Change From Baseline in New York Heart Association (NYHA) Functional Class
Description: Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea. Class II: Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea. Class III: Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea. Class IV: Unable to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: Baseline to 12 months
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Replagal® (0.2 mg/kg)
Number analyzed (Participants) | 35
participants
  Improved ≥ 1 NYHA Functional Class | 0
  Maintained NYHA Functional Class | 34
  Missing | 1

6. Secondary Outcome: Change From Baseline in Plasma Gb3
Time Frame: Baseline to 12 months
Population: ITT population. Number of participants analyzed signifies participants evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: (nmol/mL)
Arm/Group | Replagal® (0.2 mg/kg)
Number analyzed (Participants) | 34
(nmol/mL) | -1.18 (1.52)

7. Secondary Outcome: Change From Baseline in eGFR
Time Frame: Baseline to 12 months
Population: ITT population. Number of participants analyzed signifies participants evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: (mL/min/1.73m^2)
Arm/Group | Replagal® (0.2 mg/kg)
Number analyzed (Participants) | 34
(mL/min/1.73m^2) | -3.25 (10.22)

8. Secondary Outcome: Change From Baseline in Albumin/Creatinine (A/Cr) Ratio
Time Frame: Baseline to 12 months
Population: ITT population. Number of participants analyzed signifies participants evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Replagal® (0.2 mg/kg)
Number analyzed (Participants) | 34
Ratio | 178.5 (857.74)

9. Primary Outcome: Safety Evaluations
Time Frame: Baseline to 12 months
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Replagal® (0.2 mg/kg)
Number analyzed (Participants) | 35
participants
  No Adverse Event (AE) | 3
  At least one AE | 32
  At least one study drug-related AE | 2
  At least one severe or life-threatening AE | 5
  At least one Serious Adverse Event (SAE) | 6
  At least one study drug-related SAE | 0
  Discontinued due to an AE | 1
  Deaths | 1

ADVERSE EVENTS:
Time Frame: Baseline to 12 Months
Arm/Group | Replagal® (0.2 mg/kg)
Serious Adverse Events (participants affected / at risk) | 6/35
Other Adverse Events (participants affected / at risk) | 32/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Replagal® (0.2 mg/kg) (N=35)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (5)
Cardiac failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (2)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Replagal® (0.2 mg/kg) (N=35)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (3)
Dilatation atrial (Cardiac disorders) | 2 (2)
Left atrial dilatation (Cardiac disorders) | 3 (3)
Palpitations (Cardiac disorders) | 5 (6)
Hypothyroidism (Endocrine disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 7 (10)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (12)
Vomiting (Gastrointestinal disorders) | 2 (7)
Chest pain (General disorders) | 3 (4)
Oedema peripheral (General disorders) | 4 (4)
Pyrexia (General disorders) | 2 (2)
Bronchitis (Infections and infestations) | 6 (7)
Nasopharyngitis (Infections and infestations) | 10 (15)
Oral herpes (Infections and infestations) | 2 (2)
Respiratory tract infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 3 (3)
Blood glucose increased (Investigations) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 2 (3)
Electrocardiogram QT prolonged (Investigations) | 3 (3)
Troponin T increased (Investigations) | 2 (2)
Impaired fasting glucose (Metabolism and nutrition disorders) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7)
Dizziness (Nervous system disorders) | 6 (8)
Headache (Nervous system disorders) | 7 (7)
Disorientation (Psychiatric disorders) | 2 (2)
Sleep disorder (Psychiatric disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤180 days from the time submitted to Shire for review. Shire does not prohibit publication, but can require the removal of confidential information(excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication.